CLINICAL TRIAL: NCT05425030
Title: Effectiveness of a Community Health Worker-Led Low-Sodium Salt Intervention to Reduce Blood Pressure: A Cluster Randomized Controlled Trial in Rural Bangladesh
Brief Title: A Community Health Worker-Led LSSS Intervention in Bangladesh
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: BRAC University (Other); Stanford King Center for Global Development (Unknown)
Responsible Party: Principal Investigator, Pascal Geldsetzer, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 63070
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Blood Pressure; Hypertension
Keywords: Sodium; Blood Pressure; Hypertension; Low Sodium Salt Substitute; Salt Substitute; Bangladesh; Global Health; Community Health Worker
MeSH Terms: conditions — Hypertension | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The primary analysis is a cluster randomized controlled trial involving 309 households in rural Bangladesh previously identified and characterized by the BRAC James P Grant School of Public Health, BRAC University. These households will be randomly divided into three arms: (1) Control, i.e., no intervention; (2) Information only, i.e., community health workers will provide basic information on the health consequences of high blood pressure, excessive salt consumption, and feedback to the participant on the likely quantity of salt s/he consumes (estimated using a questionnaire); (3) Free LSSS Arm: The same information as in Arm 2 will be provided, but participants will receive 6 months of free low-sodium salt by delivery from the community health worker.
Who Masked: Investigator, Outcomes Assessor
Masking Description: intervention), participants cannot be blinded. Investigators not involved in the allocation and direct data collection efforts, however, including the analysts, will be blinded to which household received which intervention. Of note, the community health workers responsible for provisioning the intervention and conducting the baseline survey will be a separate team of field workers from those collecting the endline outcomes assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Free LSSS Arm (Experimental): Participants will receive 6 months of free low-sodium salt by delivery from a community health worker. In addition, the same educational information as provided in Arm 2 (Information Only Arm, below) will be provided.
  Interventions: Dietary Supplement: Low-Sodium Salt Substitute; Behavioral: Information/Education
- Information Only Arm (Active Comparator): Community health workers will provide basic information on high blood pressure, the health consequences of excessive salt consumption, and feedback to the participant on the likely quantity of salt s/he consumes (estimated using a questionnaire)
  Interventions: Behavioral: Information/Education
- No Intervention (No Intervention): Participants will not receive any intervention of any sort.

INTERVENTIONS:
Dietary Supplement: Low-Sodium Salt Substitute — Tata SuperLite low-sodium salt substitute has 30% of the weight of the product replaced with potassium chloride (KCl) which is itself a non-prescription dietary supplement. Each household randomized to the intervention arm will receive one bag (1.5kg) per month to utilize instead of their usual table/cooking salt.
  Arms: Free LSSS Arm
Behavioral: Information/Education — Community health workers will provide basic information on high blood pressure, the health consequences of excessive salt consumption, and feedback to the participant on the likely quantity of salt s/he consumes (estimated using a questionnaire)
  Arms: Free LSSS Arm; Information Only Arm

SUMMARY:
The sodium found in salt is a powerful cause of high blood pressure, and most sodium ingested by humans is from their diet. High blood pressure is known to cause heart attacks and strokes, so various public health programs have attempted to find ways for people to reduce their salt intake to avoid these complications. These programs, however, have proven challenging, as asking people to alter their food preparation practices is often met with resistance. As such, we wish to test the blood pressure-lowering effects of low sodium salt substitute (LSSS), a salt substance in which a third of the compound by weight is composed of potassium (which does not increase blood pressure) rather than sodium. Additionally, the best way of supplying LSSS to people is yet unknown. We thus propose to study the effectiveness of an LSSS product by directly providing it via community health workers in 309 households in rural Bangladesh.

DETAILED DESCRIPTION:
The overall objective of this study is to assess the effectiveness of providing access to low-sodium salt substitute (LSSS) (a compound in which a percentage of the sodium chloride (NaCl) is replaced by potassium chloride (KCl) for blood pressure (BP) reduction in a general population of adults (aged 18 years and older) in rural Bangladesh. The intervention will be delivered in the study wing by community health workers to determine if this method is an efficacious approach for blood pressure lowering in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Our target population is that of adults living in rural Bangladesh, while our study population will be comprised of adults (age ≥18 years old) living in Parbatipur, a rural/semi-rural sub-district in Dinajpur District (Rangpur Division), in the north of the country. Within Parbatipur, BRAC University has assessed 700 households for NCD risk factors as part of a larger Wellcome-trust funded multinational biobank (involving those living in Bangladesh, India, Pakistan, and Sri Lanka) to better understand the patterns and determinants of cardiovascular health in South Asian people in a cross-sectional analysis. All adults living in these surveyed households will be eligible to participate.

Exclusion Criteria:

* Exclusion criteria include subjects taking potassium-sparing diuretics, already taking potassium supplements, or those who have known kidney disease at baseline.
* All adults initially screened for intervention will undergo serum creatinine testing, with those with values >106 mMol/L for males and >97 mMol/L for female excluded from the intervention but kept in the intervention group by intention-to-treat principles to avoid breaking of randomization.
* Although minors will not be involved in the study, to avoid spillover injury to children in the intervention households, all members of intervention households under the age of 18 will also undergo urine dipstick testing. If proteinuria is detected, the household will be excluded from receiving the LSSS intervention (but followed in the intervention arm to avoid breaking randomization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure at 6 months | 6 months
  Systolic blood pressure will be treated as a continuous variable expressed in millimeters of mercury (mmHg). This measurement will be made by trained fieldworkers using Omron Series 3 automatic portable blood pressure cuffs (Omron Healthcare, Kyoto, Japan) while trial subjects are in the seated position in the left arm after 15 minutes rest. Three measurements will be taken at least 5 minutes apart to ensure accurate capture, with the mean of the second and third measurements used in the final data analysis. These measurements will be taken at both baseline (prior to the initiation of the intervention) and at the endline survey at the conclusion of the study.
Change in Diastolic Blood Pressure at 6 months | 6 months
  Diastolic blood pressure will be treated as a continuous variable expressed in millimeters of mercury (mmHg). This measurement will be made by trained fieldworkers using Omron Series 3 automatic portable blood pressure cuffs (Omron Healthcare, Kyoto, Japan) while trial subjects are in the seated position in the left arm after 15 minutes rest. Three measurements will be taken at least 5 minutes apart to ensure accurate capture, with the mean of the second and third measurements used in the final data analysis. These measurements will be taken at both baseline (prior to the initiation of the intervention) and at the endline survey at the conclusion of the study.

SECONDARY OUTCOMES:
Number of Participants with Hypertension | 6 months
  Clinical hypertension will be defined as a measured blood pressure over 140mmHg systolic or over 90mmHg diastolic (or a pre-existing diagnosis of hypertension by patient report). This outcome will be treated as a binary variable.
Number of Participants AchievingHypertension Control | 6 months
  Hypertension control will be defined as an endline survey blood pressure below 140mmHg systolic or below 90mmHg diastolic in patients previously diagnosed with hypertension or meeting our trial definition of hypertension based on the baseline survey.

CONTACTS AND LOCATIONS:
Overall Officials: Malabika Sarker, PhD, Principal Investigator — James P Grant School of Public Health, BRAC University; Pascal Geldsetzer, MD, MPH, PhD, Principal Investigator — Stanford University
Locations (1):
- BRAC University, James P Grant School of Public Health, Dhaka, Mohakhali, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang AY, Rahman M, Talukder A, Shah H, Mridha MK, Hasan M, Sarker M, Geldsetzer P. Effectiveness of a community health worker-led low-sodium salt intervention to reduce blood pressure in rural Bangladesh: protocol for a cluster randomized controlled trial. Trials. 2023 Jul 27;24(1):480. doi: 10.1186/s13063-023-07518-3. PMID 37501102